CLINICAL TRIAL: NCT05143554
Title: Efficacy of Auricular Neurostimulation for Children Adolescents and Young Adults With Chemotherapy Induced Nausea and Vomiting
Brief Title: Auricular Neurostimulation for Chemotherapy Induced Nausea and Vomiting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to accrue
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Angela Steineck, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1678523-2
Record Dates: First submitted 2021-07-06; First posted 2021-12-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: Each subject will be randomized to receive active vs sham therapy, then cross over to the other during the following cycle of chemotherapy
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active percutaneous neurostimulation (Active Comparator): Subject randomized to maximum of 5 days of active vs sham neurostimulation therapy with moderate to severe emetogenic chemotherapy admission . With the next scheduled identical chemotherapy cycle, each subject will cross over to the other one (active vs sham)
  Interventions: Device: Auricular percutaneous neurostimulation
- Sham percutaneous neurostimulation (Sham Comparator): Subject randomized to maximum of 5 days of active vs sham neurostimulation therapy with moderate to severe emetogenic chemotherapy admission . With the next scheduled identical chemotherapy cycle, each subject will cross over to the other one (active vs sham)
  Interventions: Device: Sham percutaneous neurostimulation

INTERVENTIONS:
Device: Auricular percutaneous neurostimulation — Percutaneous neurostimulation
  Other Names: IBStim
  Arms: Active percutaneous neurostimulation
Device: Sham percutaneous neurostimulation — Sham percutaneous neurostimulation
  Arms: Sham percutaneous neurostimulation

SUMMARY:
This study evaluates the efficacy of auricular percutaneous electrical nerve field stimulator in children, adolescents and young adults with chemotherapy induced nausea and vomiting.

DETAILED DESCRIPTION:
Chemotherapy induced nausea and vomiting (CINV) is a difficult to treat and potentially debilitating complication of chemotherapy. Nausea and vomiting are one of the most prevalent and problematic side effects associated with chemotherapy treatment, effecting numerous patients.

Autonomic nervous system (ANS) and the vagus nerve are important modulators of nausea and vomiting and are responsible for conveying visceral sensory information to the central nervous system responsible for nausea and vomiting. The aim of the study is to determine if stimulating a branch of the vagus nerve in the outer ear would reduce the frequency and severity of nausea and vomiting for patients undergoing chemotherapy treatment.

Subjects will be randomized to receive active vs sham (non-active) neurostimulation therapy which would be applied for maximum of 5 days at the onset of inpatient admission for moderate to severe emetogenic chemotherapy cycle. They will then cross over to the other group (active vs sham) during the admission of the following identical chemotherapy cycle. Nausea, vomiting, the need for additional antiemetic support and potential side effects will be monitored during the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are scheduled to be admitted for chemotherapy administration and who will have at least one additional cycle of the same chemotherapy
* Chemotherapy regimens must include moderate and/or severe emetogenic chemotherapy

Exclusion Criteria:

* Significant developmental delays that would prohibit participation
* Infection or severe dermatological condition of ear
* Uncontrolled or severe infection
* No implanted electrical device is permitted
* Pregnancy
* Severe cardiopulmonary disease
* Diagnosis of hemophilia or other bleeding disorders
* Diagnosis psoriasis vulgaris

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Baxter Retching Faces Scale | From the date of baseline assessment up to 7 days after completion of intervention ( day 13)
  Nausea severity assessed by pictorial nausea faces scale 0-10 (0=no nausea; 10= worse possible nausea) multiple times during hospitalization until discharge
Change in Rhodes Index of Nausea, Vomiting and Retching (INVR) | From the date of baseline assessment and during the intervention (up to day 5)
  Short 8 item questionnaire to assess severity of nausea, vomiting and retching symptoms
Assessment of Rescue Medication | From the date of baseline assessment up to 7 days after completion of intervention ~ day 13
  Number of rescue medications to be assessed on daily basis.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Wisconsin Hospital, Milwaukee, Wisconsin, United States